CLINICAL TRIAL: NCT06319859
Title: Intrathecal Non-preservative-free Morphine With Bupivacaine Versus Intrathecal Bupivacaine Alone for Analgesia in Unilateral Inguinal Hernia Repair Surgeries: A Randomized Controlled Clinical Trial.
Brief Title: Intrathecal Non-preservative-free Morphine With Bupivacaine Versus Intrathecal Bupivacaine Alone for Analgesia in Unilateral Inguinal Hernia Repair Surgeries
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, AbdElKhalik Mahmoud Shaban, Lecturer of anaesthesia, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N-72-2024
Record Dates: First submitted 2024-03-13; First posted 2024-03-20 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2024-07

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Morphine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): patients will receive 0.1 mg morphine with 15 mg heavy bupivacaine intrathecally
  Interventions: Drug: Morphine
- Group B (Active Comparator): patients will receive 15 mg heavy bupivacaine with 0.1 ml saline intrathecally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Morphine — The patients will receive 0.1 mg morphine with 15 mg heavy bupivacaine intrathecally
  Arms: Group A
Drug: Placebo — The patients will receive 15 mg heavy bupivacaine with 0.1 ml saline intrathecally
  Arms: Group B

SUMMARY:
This study will evaluate the efficacy and safety of intrathecal non-preservative-free morphine and its effect on pain in patients undergoing unilateral inguinal hernia surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-65 years old.
* Both genders.
* ASA I and II class.

Exclusion Criteria:

* Patient refusal.
* Known local anesthetic (LA) allergy.
* Skin lesions or infections at the site of needle insertion.
* Contraindications to spinal anesthesia.
* Failure of spinal anesthesia.
* ASA III and VI class.
* Central or peripheral neuropathies.
* Severe respiratory or cardiac diseases.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-08-03 (Actual); Primary Completion 2025-10-15 (Actual); Study Completion 2025-11-25 (Actual)

PRIMARY OUTCOMES:
Time to first analgesic requirement | 48 hours post-operatively
  The time to first analgesic required by the patient will be recorded

SECONDARY OUTCOMES:
Nalbuphine consumption | 48 hours post-operatively
  The amount of nalbuphine consumption as postoperative analgesia
Postoperative pain | at 2, 4,8,12,18,24,30,36,42, and 48 hours post-operatively
  Postoperative pain at rest and movement by numeric rating scale Patients will be asked to circle the number between 0 and 10, that fits best to their pain intensity. Zero represents 'no pain at all' whereas the upper limit represents 'the worst pain ever possible'
The incidence of other adverse effects | 14 days post-operatively
  The incidence of other adverse effects e.g. neurotoxicity, respiratory depression, nausea, vomiting, urine retention and pruritus will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Alaini hospital, Cairo, Egypt